CLINICAL TRIAL: NCT05892536
Title: Evaluation of the Effect of Photobiomodulation on Revascularization of Mature Non-vital Permanent Teeth Using Blood Clot as Scaffold
Brief Title: Regenerative Endodontics in Mature Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salma fathy (Other)
Responsible Party: Sponsor-Investigator, Salma fathy, Doctor of pedodontics, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 364
Record Dates: First submitted 2022-10-18; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-04

CONDITIONS: Regenerative Endodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood clot regeneration (Experimental): the regenerative procedures were performed by over-instrumentation the apices and irritating the apical tissues to induce bleeding into the root canal, then orifices plugged with MTA over blood clot and restored with GI.
  Interventions: Procedure: dental regenerative endodontics
- photo-biomodulation regeneration (Active Comparator): photobiomodulation therapy was carried out using diode laser with wavelenght 810 nm and output power 300 mW on the apical root areas of buccal and lingual surfaces at 48 hours intervals for 2 weeks after completion of the regenerative procedures which were performed by over-instrumentation the apices and irritating the apical tissues to induce bleeding into the root canal, then orifices plugged with MTA over blood clot and restored with GI.
  Interventions: Procedure: dental regenerative endodontics

INTERVENTIONS:
Procedure: dental regenerative endodontics — regenerative procedures performed in necrotic mature permanent teeth

SUMMARY:
this study was designed to compare the clinical and radiographic success of REPs after using blood clot scaffold in non-vital mature permanent teeth with or without photobiomodultion therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients free from any systemic diseases or genetic disorders.
* Children aged 9-13 years old of both sexes.
* Traumatically or cariously exposed single rooted mature permanent teeth which may be asymptomatic or manifested with dull ache pain, or spontaneous unprovoked toothache.
* Non-vital single rooted mature permanent teeth that indicated for endodontic treatment
* Swelling close to involved tooth accompanied with or without fistula.
* Negative response to cold & electrical pulp test.
* Informed Consent.

Exclusion Criteria:

* Unrestorable teeth, or that need post and core for the final restoration.
* Immature permanent teeth.
* Known allergy, sensitivity to ciprofloxacin, metronidazol.
* Uncooperativeness of child and/or parents or caregiver's behavior.
* Presence of calcific metamorphosis inside root canals.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Pulp sensibility | Every 3 months over a period of one year
  clinical evaluation of pulp sensibility using electric pulp tester as a measurement tool
Radiographic evaluation of periapical tissues | Every 3 months over a period of one year
  Radiographic evaluation using standardized digital radiograph that stored in computer for assessment of periapical tissues status using scoring system:
  1. Score 0 - No radiological changes seen compared to preoperative radiograph
  2. Score 1 - Slight decrease in radiolucency seen in periapical region
  3. Score 2 - Complete reduction or resolution of radiolucency seen in periapical region.

CONTACTS AND LOCATIONS:
Overall Officials: salma khattab, master, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No